CLINICAL TRIAL: NCT01368536
Title: A 12-week, Multi-Center, Randomized Double-Blind, Active Control Parallel Group Study to Evaluate the Efficacy and Safety of the Combination of Valturna and Amlodipine or Valturna and Chlorthalidone Versus Valturna Alone in Patients With Stage 2 Hypertension and Diabetes
Brief Title: Study to Evaluate the Efficacy and Safety of the Combination of Valturna and Amlodipine or Valturna and Chlorthalidone Versus Valturna Alone in Patients With Stage 2 Hypertension and Diabetes
Acronym: VALENCIA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Based on results from an ALTITUDE study interim analysis, testing aliskiren concomitantly with an ACE inhibitor or ARB, in diabetics with renal impairment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPV100AUS05
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension; Stage 2 Hypertension; Diabetes
Keywords: High blood pressure; diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Amlodipine; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Valturna (Experimental): At double-blind randomization, all patients received 1 tablet Valturna 150/160 mg + 1 tablet Placebo Valturna+ 1 capsule placebo for 2 weeks. From Week 2, patients received 1 tablet Valturna 150/160 mg, + 1 tablet Valturna 150/160 mg + 1 capsule placebo for 6 weeks. From Week 8, patients received 1 tablet Valturna 150/160 mg + 1 tablet Valturna 150/160 mg + 1 capsule placebo for 4 weeks.
  Interventions: Drug: Valturna; Drug: Placebo of Valturna Tablet; Drug: Placebo Capsule
- Valturna + Amlodipine (Active Comparator): At double-blind randomization, all patients received 1 tablet Valturna 150/160 mg + 1 tablet Placebo Valturna+ 1 capsule placebo for 2 weeks. From Week 2, patients received 1 tablet Valturna 150/160 mg, + 1 tablet Valturna 150/160 mg + 1 capsule 5 mg amlodipine for 6 weeks. From Week 8, patients received 1 tablet Valturna 150/160 mg + 1 tablet Valturna 150/160 mg + 1 capsule 10 mg amlodipine for 4 weeks.
  Interventions: Drug: Valturna; Drug: Amlodipine; Drug: Placebo of Valturna Tablet; Drug: Placebo Capsule
- Valturna + chlorthalidone (Active Comparator): At double-blind randomization, all patients received 1 tablet Valturna 150/160 mg + 1 tablet Placebo Valturna+ 1 capsule placebo for 2 weeks. From Week 2, patients received 1 tablet Valturna 150/160 mg, + 1 tablet Valturna 150/160 mg + 1 capsule 15 mg chlorthalidone for 6 weeks. From Week 8, patients received 1 tablet Valturna 150/160 mg + 1 tablet Valturna 150/160 mg + 1 capsule 25 mg chlorthalidonefor 4 weeks.
  Interventions: Drug: Valturna; Drug: Chlorthalidone; Drug: Placebo of Valturna Tablet; Drug: Placebo Capsule

INTERVENTIONS:
Drug: Valturna — Valturna (aliskiren 150 mg/valsartan 160 mg) tablet
Drug: Amlodipine — Amlodipine 5 mg and 10 mg capsule
  Arms: Valturna + Amlodipine
Drug: Chlorthalidone — Chlorthalidone 15 mg and 25 mg capsule
  Arms: Valturna + chlorthalidone
Drug: Placebo of Valturna Tablet — Matching placebo of valturna tablet
Drug: Placebo Capsule — Matching placebo of Amlodipine capsule OR Matching placebo of chlorthalidone capsule

SUMMARY:
This was a study to assess the safety and efficacy of Valturna and amlodipine or Valturna and chlorthalidone when compared to Valturna alone in patients with stage 2 hypertension and diabetes mellitus 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 2 hypertension within protocol limits at randomization
* Patients with type 2 diabetes mellitus with HgA1c less than or equal to 9%
* Patients with newly diagnosed hypertension or patients who have not received antihypertensive therapy for at least 4 weeks prior to screening

Exclusion Criteria:

* Patients taking 4 or more antihypertensive medications at screening visit
* Patients with uncontrolled BP (> 140/90 mmHg) while taking 3 or more antihypertensives at their maximum approved doses
* Type 2 diabetes mellitus requiring insulin treatment
* Patients with HgA1c > 9%
* Patients with known gout
* Known history of cancer within the past 5 years
* Patients who are pregnant or nursing mothers
* Patients who have participated in an investigational clinical trial within the 30 days prior to screening.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (83):
- United States (81):
  - Novartis Investigative Site, Athens, Alabama
  - Novartis Investigative Site, Florence, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Montgomery, Alabama
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Buena Park, California
  - Novartis Investigative Site, Fair Oaks, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Healdsburg, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orangevale, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Roseville, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, West Covina, California
  - Novartis Investigative Site, Shelton, Connecticut
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Lauderdale Lakes, Florida
  - Novartis Investigative Site, North Miami Beach, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Gurnee, Illinois
  - Novartis Investigative Site, Lansing, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Beltsville, Maine
  - Novartis Investigative Site, Waltham, Massachusetts
  - Novartis Investigative Site, Wellesley Hills, Massachusetts
  - Novartis Investigative Site, Brooklyn Center, Minnesota
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Ozark, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Trenton, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Camillus, New York
  - Novartis Investigative Site, Asheboro, North Carolina
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Lyndhurst, Ohio
  - Novartis Investigative Site, Zanesville, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Reading, Pennsylvania
  - Novartis Investigative Site, Uniontown, Pennsylvania
  - Novartis Investigative Site, Wallingford, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Easley, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Fayetteville, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lake Jackson, Texas
  - Novartis Investigative Site, Pasadena, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Richardson, Texas
  - Novartis Investigative Site, St. George, Utah
  - Novartis Investigative Site, Arlington, Virginia
- Puerto Rico (2):
  - Novartis Investigative Site, Carolina
  - Novartis Investigative Site, San Juan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 975 patients screened, 417 were randomized.
Period: Overall Study
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone
Started | 138 | 137 | 142
Full Analysis Set | 138 | 137 | 141 (One patient was excluded from efficacy analysis as there was no post baseline data)
Completed | 87 | 78 | 83
Not Completed | 51 | 59 | 59
Not completed — Adverse Event | 5 | 6 | 8
Not completed — Abnormal laboratory value(s) | 0 | 1 | 2
Not completed — Abnormal test procedure result(s) | 0 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 7 | 2 | 2
Not completed — No longer required study medication | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5 | 4
Not completed — Lost to Follow-up | 3 | 3 | 5
Not completed — Administrative problems | 34 | 39 | 35
Not completed — Protocol deviation | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone | Total
Number analyzed (Participants) | 138 | 137 | 141 | 416
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (8.65) | 56.0 (9.56) | 54.6 (9.35) | 55.1 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 73 | 70 | 216
  Male | 65 | 64 | 71 | 200

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) After 12 Weeks of Treatment Ending With the Combination of Valturna and Amlodipine Versus Valturna Alone
Description: Sitting BP was measured at trough (24 hours ± 3 hours postdose) and recorded at all study visits. At the first study visit, the patient had his/her BP measured in both arms; the arm in which the highest sitting DBP was found was used for all subsequent readings throughout the study. At each study visit, after the patient had been sitting for 5 minutes, SBP were measured 3 times using a standard mercury sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1- to 2-minute intervals and the mean of those 3 measurements was used as the average sitting office BP for that visit.
Time Frame: Baseline, 12 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Valturna | Valturna + Amlodipine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in MSSBP After 12 Weeks of Treatment Ending With Between the Valturna + Chlorthalidone Combination and Valturna Alone
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Valturna | Valturna + Chlorthalidone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) After 12 Weeks of Treatment
Description: Sitting blood pressure (BP) was measured at trough (24 hours ± 3 hours postdose) and recorded at all study visits. At the first study visit, the patient had his/her BP measured in both arms; the arm in which the highest sitting DBP was found was used for all subsequent readings throughout the study. At each study visit, after the patient had been sitting for 5 minutes, DBP were measured 3 times using a standard mercury sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1- to 2-minute intervals and the mean of those 3 measurements was used as the average sitting office BP for that visit.
Time Frame: Baseline, 12 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Responders After Treatment
Description: Responders are defined as patients with MSSBP <130 mmHg or a decrease from baseline in MSSBP of ≥20 mmHg
Time Frame: Baseline, 12 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control After Treatment
Description: Patient with blood pressure control is defined as patients achieving MSSBP <130 mmHg and MSDBP <80 mmHg.
Time Frame: 12 weeks
Population: The study was terminated and consequentially was underpowered for adequate statistical analysis
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death to Assess Safety and Tolerability of Treatment With Valturna and Chlorthalidone or Valturna and Amlodipine Versus Valturna Alone
Time Frame: 12 weeks
Population: Safety Set - Consists of all patients who received at least one dose of the double-blind study drug. Patients were analyzed according to the treatment that they received.
Measure: Number; unit: Participants
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone
Number analyzed (Participants) | 138 | 137 | 142
Participants
  Adverse Events | 62 | 54 | 58
  Serious Adverse Events | 0 | 0 | 0
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Valturna | Valturna + Amlodipine | Valturna + Chlorthalidone
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/137 | 0/142
Other Adverse Events (participants affected / at risk) | 23/138 | 16/137 | 23/142
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valturna (N=138) | Valturna + Amlodipine (N=137) | Valturna + Chlorthalidone (N=142)
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 2
Dizziness (Nervous system disorders) | 3 | 4 | 11
Headache (Nervous system disorders) | 16 | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.